CLINICAL TRIAL: NCT07114393
Title: Optimization of Complex Percutaneous Coronary Intervention With Liberal Use of Intracoronary Imaging Versus Contemporary Practice
Acronym: OPTIMIZE-PCI 2
Status: Recruiting | Type: Observational
Sponsor: Cathreine BV (Other)
Collaborators: Philips Healthcare (Industry); Boston Scientific Corporation (Industry); Abbott Medical Devices (Industry); Salveo Diagnostics (Industry)
Responsible Party: Principal Investigator, Koen Teeuwen, MD PhD, Cathreine BV
Other Study IDs: CathreineBV-OP2
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease; Coronary Artery Disease (Left Main); Chronic Total Occlusion (CTO); Bifurcation Coronary Artery Disease
Keywords: percutaneous coronary intervention; intracoronary imaging; stent optimization; complex coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-implementation cohort: This group will serve as the control cohort before implementation of a new intracoronary imaging protocol. Data from the national PCI registry, which will be supplemented with an additional set of procedural variables. Data on the percentage of use of intracoronary imaging in complex coronary lesions by the individual interventional cardiologist will be collected. This will establish a benchmark from which individual interventional cardiologists must increase their use of intracoronary imaging. This will be the pre-implementation cohort that will be used as the comparator in the final evaluation.
- Post-implementation cohort: This is the cohort in which a new intracoronary imaging protocol will be implemented. Main goal of this protocol is the increase the use of intracoronary imaging during complex PCI in the Netherlands. The duration of this phase will be approximately 1-2 year.
  Interventions: Behavioral: Liberal use of intracoronary imaging during complex PCI

INTERVENTIONS:
Behavioral: Liberal use of intracoronary imaging during complex PCI — A new protocol regarding use of intracoronary imaging will be implemented in multiple PCI centers in the Netherlands. Main goal of this protocol will be to increase the use of imaging in complex PCI in the Netherlands. Moreover operators will be trained according to the new protocol and on site training will be organized to improve the skills in using imaging during complex PCI.Operators are requested to use of intracoronary imaging preferentially in all complex coronary lesions, but at least increase their use with at least 50% and minimum of 25% of the cases. Throughout the second phase, individual participating operators will receive personalized feedback on their use of intracoronary imaging at multiple intervals. Based on this result, the implementation process will be refined as necessary. These intermediate measurements will also be shared with all participating centres anonymous.
  Groups: Post-implementation cohort

SUMMARY:
Coronary artery disease remains a leading cause of mortality worldwide and is commonly treated with percutaneous coronary intervention (PCI). Typically, PCI is guided by invasive coronary angiography (ICA). However, ICA has inherent limitations in accurately assessing vessel dimensions, calcium burden, circumferential tissue and whether a stent has achieved full expansion. [1] Therefore ICA alone is insufficient for guiding stent optimization, especially in complex lesions which are most vulnerable to long-term stent failure. [2] To overcome the limitations of ICA, intracoronary imaging can be used to guide and optimize PCI. The advantages of intracoronary imaging include obtaining larger lumen areas, better stent expansion and strut apposition, full lesion stent coverage and identifying stent complications. Multiple randomized studies have shown that these advantages translate into a reduction in major adverse cardiovascular events (MACE) in complex PCI. Consequently, the recommendation for intracoronary imaging has been upgraded in the most recent guidelines. [3-6] Despite robust evidence supporting its benefits, intracoronary imaging remains relatively underused in real-world practice and in the Netherlands it is only used in 7% of complex PCI procedures. [7] This underutilization may be attributed to several factors, including operator and hospital-dependent issues such as lack of experience, reluctance to spend additional time on intracoronary imaging and concerns about its cost-effectiveness. [8] Therefore, initiating an implementation project to incorporate intracoronary imaging into routine use in the catheterization lab during complex PCI would be highly valuable. [9] Such a project could make imaging-guided PCI the standard of care in complex PCI. Additionally, it could evaluate the cost-effectiveness of routine intracoronary imaging during complex PCI.

For this reason we designed the OPTIMIZE-PCI II, a national registry-based quality improvement project. This project is aimed at implementing a liberal intracoronary imaging-guided strategy for complex PCI across multiple centres in the Netherlands, with data extraction from the Netherlands Heart Registration (NHR) database. The objective of the OPTIMIZE-PCI II is to establish a routine use of intracoronary imaging in complex PCI, to determine if this approach reduces adverse cardiac events in real-world practice, and evaluate its cost-effectiveness.

DETAILED DESCRIPTION:
Design and outcomes measures will be discusses elsewhere. Additional information: Patients in this observational, registry study, will be included by the Netherlands heart registration (NHR). The NHR is an independent organization in which Dutch hospitals prospectively register standard sets of baseline, procedural and outcome data for all invasive cardiac procedures, including PCI. Data provided to the NHR are extensively checked on completeness and quality, reviewed with audit reports by independent trained research nurses and discussed by cardiologists in registration committees. Multiple audits are conducted annually by the NHR for data validation and verification. A waiver for informed consent for analysis with the data of the NHR data registry is obtained.

This study will be a quality improvement project.

ELIGIBILITY:
Inclusion Criteria:

All patients above the age of 18, included in the Netherlands Heart Registration (NHR) quality database after receiving PCI in complex coronary lesions, will be included in the analyses of this project.

Complex lesions include:

Left main A stenosis of >50% and/or a FFR ≤ 0.80 and iFR ≤ 0.89 in the left main.

Severely calcified lesion Defined as use of calcium modification therapy (e.g. cutting balloon, scoring balloon, rotablation, orbital atherectomy, intravascular lithotripsy).

Chronic total occlusion

Coronary CTO is defined as an obstruction of the coronary artery with the following classic lesion characteristics:

* TIMI flow 0
* Absence of contrast stasis at the site of the proximal capillaries
* Presence of collateral vessels
* Estimated occlusion duration of at least 3 months.

Ostial lesion Lesion at the origin (within 5 mm) of a major coronary vessel (LM, LAD, RCX and RCA).

Severely calcified lesion. Long lesion A vessel treated with one or multiple stents with a total stent length of ≥38 mm is considered a long lesion.

Bifurcation (true) A coronary artery narrowing occurring adjacent to, and/or involving, the origin of a significant side branch ≥ 2.5mm. Only true bifurcation will be included, i.e. medina 1,1,1/1,0,1/0,1,1.

In-stent restenosis A reduction ≥50% of the luminal diameter within the previously stented segment or the vessel segments 5 mm proximal and distal to the stent (the "stent edges"), as assessed by coronary angiography.

Exclusion Criteria:

* Non complex PCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population exists of patients registered in our national PCI registration of the Netherlands Heart Registration after receiving complex PCI. All indications are included (ACS and non-ACS, OHCA, cardiogenic shock).
Sampling Method: Non-Probability Sample
Enrollment: 11092 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of target vessel revascularization, myocardial infarction and all-cause mortality | 1 year
  The primary composite end point of major adverse cardiac events is the occurrence of target vessel revascularization, myocardial infarction and all-cause mortality.

SECONDARY OUTCOMES:
Occurrence of all cause mortality | 30 days, 1 year
  all cause mortality, confirmed by verifying the vital status of a patient in the Personal Records Database.
Occurrence of target vessel revascularization | 30 days and 1 year
  Target vessel revascularization, defined as a revascularization by percutaneous coronary intervention or coronary artery bypass grafting in the same vessel(s) that had been treated at the index procedure, excluding staged procedures.
Occurrence of myocardial infarction | 30 days 1 year
  Myocardial infarction, defined as an increase and/or decrease in one or more cardiac biomarkers by at least one value above the 99th percentile of the upper limit where at least one of the following symptoms is present: 1) symptoms appropriate to ischemia, 2) new significant ST-segment or T-wave abnormalities or bundle branch block, 3) development of pathological Q-waves on the electrocardiogram (ECG), 4) imaging demonstrated new loss of viable myocardial tissue or new wall motion abnormalities, 5) identification of intracoronary thrombus on angiography or autopsy.
Occurrence of stent thrombosis | 30 days, 1 year
  Defined as angiographically or pathologically confirmed thrombus within the stent or within 5 mm proximal or distal to the stent, occurring within 1 year, with at least one of the following criteria present within 48 hours:
  Acute onset of ischemic symptoms at rest
  New ischemic ECG changes suggestive of acute ischemia
  Characteristic rise or fall in cardiac biomarkers
  Occlusive thrombus (TIMI flow grade 0 or 1)
  Non-occlusive, visibly present thrombus (angiographically confirmed)
Occurrence of target lesion revascularization | 30 days, 1 year
  defined as a unplanned revascularization by percutaneous coronary intervention or coronary artery bypass grafting in a lesion <5 mm distally or proximally of the lesion that had been treated at the index procedure, excluding staged procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina hospital Eindhoven, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Koskinas KC, Nakamura M, Raber L, Colleran R, Kadota K, Capodanno D, Wijns W, Akasaka T, Valgimigli M, Guagliumi G, Windecker S, Byrne RA. Current use of intracoronary imaging in interventional practice - Results of a European Association of Percutaneous Cardiovascular Interventions (EAPCI) and Japanese Association of Cardiovascular Interventions and Therapeutics (CVIT) Clinical Practice Survey. EuroIntervention. 2018 Jul 20;14(4):e475-e484. doi: 10.4244/EIJY18M03_01. PMID 29537966
- [Background] Bresnahan JF, Kitchell BB, Wildman MF. Facial hair barbering in rats. Lab Anim Sci. 1983 Jun;33(3):290-1. PMID 6876735
- [Background] Stone GW, Christiansen EH, Ali ZA, Andreasen LN, Maehara A, Ahmad Y, Landmesser U, Holm NR. Intravascular imaging-guided coronary drug-eluting stent implantation: an updated network meta-analysis. Lancet. 2024 Mar 2;403(10429):824-837. doi: 10.1016/S0140-6736(23)02454-6. Epub 2024 Feb 21. PMID 38401549
- [Background] van Beek KAJ, Timmermans MJC, Derks L, Cheng JM, Kraaijeveld AO, Arkenbout EK, Schotborgh CE, Brouwer J, Claessen BE, Lipsic E, Polad J, van Nunen LX, Sjauw K, van Veghel D, Tonino PA, Teeuwen K; 'on behalf of the PCI registration committee of The Netherlands Heart Registration'. Contemporary Use of Post-Dilatation for Stent Optimization During Percutaneous Coronary Intervention; Results From the Netherlands Heart Registration. Catheter Cardiovasc Interv. 2025 Mar;105(4):870-877. doi: 10.1002/ccd.31404. Epub 2025 Jan 8. PMID 39777867